CLINICAL TRIAL: NCT01607450
Title: Modulation of Human Myocardial Metabolism by GLP-1 Dose Response
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1010002497; R21HL092799 (NIH)
Record Dates: First submitted 2012-05-21; First posted 2012-05-30 (Estimated); Results first posted 2016-02-17 (Estimated); Last update posted 2016-02-17 (Estimated); Status verified 2016-01

CONDITIONS: Type 2 Diabetes Mellitus; Healthy
Keywords: Type 2 diabetes mellitus; lean healthy control
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Glucagon-Like Peptide 1; Sodium Chloride; Saline Solution

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Saline (Other): 12 hour saline (control) infusion prior to PET study
  Interventions: Drug: Saline
- GLP-1 Low dose (Experimental): GLP-1 Low Dose: 0.5 pmol/kg/min for 12 hours prior to PET study
  Interventions: Drug: GLP-1 Low Dose
- GLP-1 Mid-Range Dose (Experimental): GLP-1 Mid-Range Dose: 1.5 pmol/kg/min for 12 hours prior to PET study
  Interventions: Drug: GLP-1 Mid-Range Dose
- GLP-1 High Dose (Experimental): GLP-1 High Dose: 4.0 pmol/kg/min for 12 hours prior to PET study
  Interventions: Drug: GLP-1 High Dose

INTERVENTIONS:
Drug: GLP-1 Low Dose — 0.5mmol/kg/hr GLP-1 for 12 hours prior to PET study
  Arms: GLP-1 Low dose
Drug: GLP-1 Mid-Range Dose — 1.5mmol/kg/min for 12 hours prior to PET study
  Arms: GLP-1 Mid-Range Dose
Drug: GLP-1 High Dose — 4.0mmol/kg/min GLP-1 for 12 hours prior to PET study
  Arms: GLP-1 High Dose
Drug: Saline — Normal saline placebo infusion for 12 hours prior to PET study
  Other Names: Normal Saline
  Arms: Saline

SUMMARY:
The objective of this proposal is to provide quantitative dose-response data for effects of GLP-1 on myocardial glucose uptake in healthy control subjects and obese type 2 diabetic subjects, in support of the design of later studies evaluating therapeutic applications of GLP-1 to heart disease.

Aim 1: To measure the effects of GLP-1 infusion on myocardial fuel selection in lean healthy humans under fasting (fatty acid-dominant) conditions. Four groups of 10 lean healthy subjects will be studied during infusions of 0 (saline control), 0.5, 1.5, and 4.0 pmol/kg/min GLP-1 (one study per subject). Cardiac metabolism will be measured using PET, using a dual-tracer approach which allows measurement of myocardial glucose uptake (the primary endpoint) along with total oxidation rate and myocardial perfusion (secondary endpoints). In concert with measures of circulating metabolites and regulatory hormones, the investigators will produce the most comprehensive assessment of actions of GLP-1 on myocardial metabolism in humans to date. Effects of each dose will be compared to the saline control, plus the investigators will combine all data and use nonlinear curve-fitting to derive sensitivity (ED50) and maximal responses for GLP-1 effects on myocardial glucose uptake.

Aim 2: To measure the effects of GLP-1 infusion on myocardial fuel selection in obese type 2 diabetic humans under fasting (fatty acid-dominant) conditions Four groups of 10 obese type 2 diabetic subjects will be studied during infusions of 0, 0.5, 1.5, and 4.0 pmol/kg/min GLP-1 as under Aim 1. Analyses will be parallel to those described under Aim 1. Results from Aims 1 and 2 will be combined to allow direct comparison of the dose-response between nondiabetic control and type 2 diabetic subjects.

No literature has been published to inform dose selection in the design of clinical trials of GLP-1 for modulation of heart fuel selection. With our expertise and experience in PET measurement of heart metabolism in diabetes, the investigators are uniquely positioned to fill this gap in knowledge. These studies are a necessary preamble to further evaluation of the potential for GLP-1 based treatments in heart disease.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-60
* Lean subjects will be defined as having a BMI <25 kg/m2, in good general health, taking no regular medications
* Diabetic subjects will be obese (BMI >30 kg/m2 but <40 kg/m2), HbA1c 7.0-10.0%, treated with diet and exercise plus oral agents or injected insulin. All diabetic subjects will be treated with injected insulin for 2 weeks prior to study, to avoid potential confounding effects of other antidiabetic agents.

Exclusion Criteria:

* Chronic illnesses or infections (other than type 2 diabetes)
* Known coronary artery disease or abnormal ECG on screening evaluation
* Blood pressure > 160/100 mmHg on two occasions during screening evaluations. Current use of 3 or fewer blood pressure medications with blood pressure below this cutpoint will be acceptable.
* Total cholesterol > 240 mg/dL. Current use of 2 or fewer lipid lowering agents with cholesterol below this cutpoint will be acceptable.
* Diabetic subjects: Treatment with a GLP-1 agonist or DPP4 inhibitor within the past 6 months
* Known intolerance to injected GLP-1 agonist
* Treatment with PPAR gamma agonists currently or within the past 6 months
* Recognized microvascular complications (retinopathy, nephropathy, neuropathy)
* Unwillingness or inability to use injected insulin for the purposes of this study
* Chronic pain or other physical conditions which limit ability to remain supine for the duration of the study protocol
* History of claustrophobia, musculoskeletal or other factors which would result in an inability to comfortably remain within PET scanner gantry for the duration of the imaging protocol
* Occupational, investigational or other known radiation exposure which, together with the planned radiologic studies, will result in greater than 500 mrem total exposure in a contiguous 12 month period
* For female participants, current pregnancy

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2010-05; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kieren J Mather, MD, Principal Investigator — Indiana University
Locations (1):
- Indiana Clinical Research Center, Indianapolis, Indiana, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Lean Placebo: 12 hour placebo (saline) infusion prior to PET study
  Placebo: Saline placebo infusion for 12 hours prior to PET study
- Lean GLP-1 Mid-Range Dose; Type 2 DM GLP-1 Mid-Range Dose: GLP-1 Mid-Range Dose: 1.5 pmol/kg/min for 12 hours prior to PET study
- Lean GLP-1 Low Dose; Type 2 DM GLP-1 Low Dose: GLP-1 Low Dose: 0.5 pmol/kg/min for 12 hours prior to PET study
- Lean GLP-1 High Dose: GLP-1 High Dose: 4.0 pmol/kg/min for 12 hours prior to PET study
- Type 2 DM GLP-1 High Dose: GLP-1 High Dose: 1.5 pmol/kg/min for 12 hours prior to PET study
Period: Overall Study
Arm/Group | Lean Placebo | Lean GLP-1 Mid-Range Dose | Type 2 DM GLP-1 Mid-Range Dose | Lean GLP-1 Low Dose | Type 2 DM GLP-1 Low Dose | Lean GLP-1 High Dose | Type 2 DM GLP-1 High Dose
Started | 6 | 8 | 7 | 11 | 1 | 0 | 0
Completed | 6 | 8 | 7 | 11 | 1 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Lean Saline: 12 hour placebo (saline) infusion prior to PET study
  Placebo: Saline placebo infusion for 12 hours prior to PET study
- Lean GLP-1 0.5 Pmol/kg/Min; Type 2 DM GLP-1 0.5 Pmol/kg/Min: GLP-1 Low Dose: 0.5 pmol/kg/min for 12 hours prior to PET study
- Lean GLP-1 1.5 Pmol/kg/Min; Type 2 DM GLP-1 1.5 Pmol/kg/Min: GLP-1 Mid-Range Dose: 1.5 pmol/kg/min for 12 hours prior to PET study
- Lean GLP-1 4.0 Pmol/kg/Min; Type 2 DM GLP-1 4.0 Pmol/kg/Min: GLP-1 High Dose:4.0 pmol/kg/min for 12 hours prior to PET study
- Total: Total of all reporting groups
Arm/Group | Lean Saline | Lean GLP-1 0.5 Pmol/kg/Min | Type 2 DM GLP-1 0.5 Pmol/kg/Min | Lean GLP-1 1.5 Pmol/kg/Min | Type 2 DM GLP-1 1.5 Pmol/kg/Min | Lean GLP-1 4.0 Pmol/kg/Min | Type 2 DM GLP-1 4.0 Pmol/kg/Min | Total
Number analyzed (Participants) | 6 | 11 | 1 | 8 | 7 | 0 | 0 | 33
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.5 (10.6) | 38.0 (6.0) | 42 (0) | 46.0 (5.8) | 45.1 (7.9) |  |  | 42.7 (7.9)
Gender [Number; unit: participants]
  Female | 5 | 3 | 0 | 3 | 1 |  |  | 12
  Male | 1 | 8 | 1 | 5 | 6 |  |  | 21
Region of Enrollment [Number; unit: participants]
  United States | 6 | 11 | 1 | 8 | 7 |  |  | 33
Body Mass Index (kg/m2) [Mean (Standard Deviation); unit: kg/m^2] | 23.9 (1.6) | 23.0 (1.5) | 31.0 (0) | 22.9 (1.8) | 30.3 (1.7) |  |  | 25.7 (1.7)
HbA1c (%) [Mean (Standard Deviation); unit: %] | 5.47 (0.40) | 5.47 (0.40) | 7.0 (0) | 5.56 (0.34) | 8.40 (3.02) |  |  | 6.48 (1.24)

OUTCOME MEASURES:

1. Primary Outcome: Myocardial Glucose Uptake.
Description: Myocardial glucose uptake measured using 18FDG PET, quantified using a 3-compartment model with a lumped constant of 1.0.
Time Frame: After 12 hours of glucagon-like peptide 1 (GLP-1) exposure
Measure: Mean (Standard Deviation); unit: umol/min/100g
Groups:
- Type 2DM GLP-1 1.5 Pmol/kg/Min: GLP-1 Mid-Range Dose: 1.5 pmol/kg/min for 12 hours prior to PET study
- Type 2 DM GLP-1 High Dose: GLP-1 High Dose: 4.0 pmol/kg/min for 12 hours prior to PET study
Arm/Group | Lean Saline | Lean GLP-1 Low Dose | Type 2 DM GLP-1 Low Dose | Lean GLP-1 1.5 Pmol/kg/Min | Type 2DM GLP-1 1.5 Pmol/kg/Min | Lean GLP-1 High Dose | Type 2 DM GLP-1 High Dose
Number analyzed (Participants) | 6 | 11 | 1 | 8 | 7 | 0 | 0
umol/min/100g | 7.46 (8.49) | 7.22 (9.26) | 0.05 (0) | 20.89 (12.47) | 5.57 (19.39) |  |

2. Secondary Outcome: Myocardial Blood Flow
Description: Myocardial perfusion derived from acetate kinetics
Time Frame: After 12 hours of GLP-1 exposure
Measure: Mean (Standard Deviation); unit: ml/min/100g
Arm/Group | Lean Saline | Lean GLP-1 Low Dose | Type 2 DM GLP-1 Low Dose | Lean GLP-1 1.5 Pmol/kg/Min | Type 2DM GLP-1 1.5 Pmol/kg/Min | Lean GLP-1 High Dose | Type 2 DM GLP-1 High Dose
Number analyzed (Participants) | 6 | 11 | 1 | 8 | 7 | 0 | 0
ml/min/100g | 34.66 (4.60) | 44.44 (9.17) | 47.61 (0) | 35.30 (7.35) | 51.19 (19.39) |  |

3. Secondary Outcome: Myocardial Total Oxidation Rate
Description: MVO2 derived from acetate kinetics
Time Frame: After 12 hours of GLP-1 exposure
Measure: Mean (Standard Deviation); unit: ml/min/100g
Arm/Group | Lean Saline | Lean GLP-1 Low Dose | Type 2 DM GLP-1 Low Dose | Lean GLP-1 1.5 Pmol/kg/Min | Type 2DM GLP-1 1.5 Pmol/kg/Min | Lean GLP-1 High Dose | Type 2 DM GLP-1 High Dose
Number analyzed (Participants) | 6 | 11 | 1 | 8 | 7 | 0 | 0
ml/min/100g | 15.25 (2.39) | 30.21 (14.32) | 65.30 (0) | 18.57 (3.78) | 59.85 (30.47) |  |

4. Secondary Outcome: Cardiac Index
Description: Impedance cardiography-derived measurement of cardiac index, assessed following 12 hour exposure to treatment condition concurrent with the PET measurements.
Time Frame: After 12 hours of GLP-1 exposure
Population: Analyses performed only on the groups with relevant primary outcome data observed
Measure: Mean (Standard Deviation); unit: L/min/m^2
Arm/Group | Lean Saline | Lean GLP-1 0.5 Pmol/kg/Min | Type 2 DM GLP-1 0.5 Pmol/kg/Min | Lean GLP-1 1.5 Pmol/kg/Min | Type 2 DM GLP-1 1.5 Pmol/kg/Min | Lean GLP-1 4.0 Pmol/kg/Min | Type 2 DM GLP-1 4.0 Pmol/kg/Min
Number analyzed (Participants) | 6 | 0 | 0 | 8 | 7 | 0 | 0
L/min/m^2 | 3.00 (0.52) |  |  | 2.88 (0.31) | 2.90 (0.51) |  |

5. Secondary Outcome: GLP-1 Concentrations
Description: Achieved GLP-1 concentrations at the end of the 12 hour treatment exposure
Time Frame: After 12 hours of GLP-1 exposure
Population: Analyses performed only on the groups with relevant primary outcome data observed
Measure: Mean (Standard Deviation); unit: pmol/L
Arm/Group | Lean Saline | Lean GLP-1 0.5 Pmol/kg/Min | Type 2 DM GLP-1 0.5 Pmol/kg/Min | Lean GLP-1 1.5 Pmol/kg/Min | Type 2 DM GLP-1 1.5 Pmol/kg/Min | Lean GLP-1 4.0 Pmol/kg/Min | Type 2 DM GLP-1 4.0 Pmol/kg/Min
Number analyzed (Participants) | 6 | 0 | 0 | 8 | 7 | 0 | 0
pmol/L | 61.7 (33.5) |  |  | 302.1 (149.1) | 307.8 (86.2) |  |

ADVERSE EVENTS:
Groups:
- Lean GLP-1 4.0 Pmol/kg/Min; Type 2 DM GLP-1 4.0 Pmol/kg/Min: GLP-1 High Dose: 4.0 pmol/kg/min for 12 hours prior to PET study
Arm/Group | Lean Saline | Lean GLP-1 0.5 Pmol/kg/Min | Type 2 DM GLP-1 0.5 Pmol/kg/Min | Lean GLP-1 1.5 Pmol/kg/Min | Type 2 DM GLP-1 1.5 Pmol/kg/Min | Lean GLP-1 4.0 Pmol/kg/Min | Type 2 DM GLP-1 4.0 Pmol/kg/Min
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/11 | 0/1 | 0/8 | 0/7 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/6 | 1/11 | 0/1 | 0/8 | 0/7 | 0/0 | 0/0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lean Saline (N=6) | Lean GLP-1 0.5 Pmol/kg/Min (N=11) | Type 2 DM GLP-1 0.5 Pmol/kg/Min (N=1) | Lean GLP-1 1.5 Pmol/kg/Min (N=8) | Type 2 DM GLP-1 1.5 Pmol/kg/Min (N=7) | Lean GLP-1 4.0 Pmol/kg/Min (N=0) | Type 2 DM GLP-1 4.0 Pmol/kg/Min (N=0)
Nausea (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Nausea associated with the infusion of GLP-1

LIMITATIONS AND CAVEATS:
This was a dose-finding study of myocardial responses to systemically infused GLP-1. After ascertaining no detectable response in controls with low dose, we completed mid dose studies. Finding an important difference there we did not do the high dose

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No